CLINICAL TRIAL: NCT00329732
Title: Double-Blind, Placebo Controlled Trial Of Greater Occipital Nerve Block For The Treatment Of Migraine Status
Brief Title: Research Study of Greater Occipital Nerve Block As A Treatment For Prolonged Migraine Attacks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to inadequate recruitment
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Bruce Smith, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GON-DBPC/WBY
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lidocaine/Bupivicaine (Active Comparator)
  Interventions: Drug: 0.5% bupivicaine and 2% lidocaine
- saline (Placebo Comparator): matching volume of saline injected
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: 0.5% bupivicaine and 2% lidocaine — The injectors will infiltrate an area of 2cm along the occipital ridge centering around the occipital artery or around the site 1/3 from the mastoid to the inion. If the subject has a bilateral headache or the headache is known to switch sides then the block will be performed bilaterally. If the headache is strictly unilateral, the block will be performed only on the side of the headache
  Arms: Lidocaine/Bupivicaine
Drug: Saline placebo — matching volume of saline (placebo)
  Arms: saline

SUMMARY:
Greater Occipital Nerve Blocks (GONB) are a common procedure used for the treatment of headache. The GONB procedure involves a series of injections into the greater occipital nerve (a spinal nerve located at the back of your head). The purpose of this study is to determine whether GONB is effective for the treatment of prolonged migraine attacks. This study is placebo controlled, which means that half of the patients participating will receive injections of active study drug (lidocaine plus bupivicaine) and half of the patients will receive injections of saline (placebo). The study is also blinded which means that neither you nor the study staff will know whether you received active study drug or placebo. The study remains blinded only for the first 30 minutes, at which point additional treatments (including GONB) can be administered at the discretion of your treating physician.

40 patients are expected to participate in this research study. This study is being conducted at Thomas Jefferson University only.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, male or female, between the ages of 18 and 80 years old (inclusive) with a previous diagnosis fulfilling IHS criteria for episodic migraine
* Presenting to clinic in migraine status, meaning the migraine has continued for greater than or equal to 3 days but less than 3 months.
* Pain must be reported as at least moderate pain level at time of injections

Exclusion Criteria:

A subject is ineligible to participate in this study if he/she satisfies any of the following criteria:

* Subjects who have received greater occipital nerve blocks in the past
* Subjects who in their own or the investigator's opinion are unable to describe their symptoms
* Subjects who are pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Young, M.D., Principal Investigator — Jefferson Headache Center
Locations (1):
- Jefferson Headache Center/Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine/Bupivicaine | Saline (Placebo)
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine/Bupivicaine | Saline (Placebo) | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 2 |  | 2
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Experiencing Significant Change on a 4 Point Pain Scale at 30 Minutes Post-injection, Active Drug Versus Placebo. Significant Change is Defined as a Change on the 4 Point Pain Scale From Moderate or Severe to Mild. No Pain Equals 0.
Time Frame: 30 minutes
Population: No analysis was done. Study was terminated.
Arm/Group | Lidocaine/Bupivicaine
Number analyzed (Participants) | 0

2. Secondary Outcome: Secondary Measures Include:Percentage of Subjects Achieving a Significant Change on a 10 Point Pain Scale at 30 Minutes Post-injection, Active Drug Versus Placebo;
Time Frame: 30 minutes
Reporting Status: Not Posted
Measure: Number; unit: participants

3. Secondary Outcome: Percentage of Subjects Achieving a Significant Change on a 100mm Visual Analogue Scale (VAS) at 30 Minutes Post-injection, Active Drug Versus Placebo. Significant Change is Defined as a Greater Than or Equal to 2cm Change.
Time Frame: 30 minutes
Reporting Status: Not Posted
Measure: Number; unit: participants

4. Secondary Outcome: Percentage of Subjects Achieving Resolution of Associated Symptoms of Nausea, Vomiting, Photophobia, Phonophobia, Osmophobia, Allodynia Measured During the First 30 Minutes Post-injection, Active Drug Versus Placebo;
Time Frame: 30 minutes
Reporting Status: Not Posted
Measure: Number; unit: participant

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Lidocaine/Bupivicaine | Saline (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes